CLINICAL TRIAL: NCT03566628
Title: Post-anaesthetic Shivering Amongst Patients Undergoing Cerebral Angiography: A Randomised Trial
Brief Title: Post-anaesthetic Shivering Amongst Patients Undergoing Cerebral Angiography
Acronym: SHIVERS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Hospital Carlos Van Buren (Other)
Responsible Party: Principal Investigator, Nathalie Lopez, Principal Investigator, Universidad de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UV-002
Record Dates: First submitted 2018-05-27; First posted 2018-06-25 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Cerebral Angiography; Shivering
Keywords: Cerebral Angiography; Shivering; Anaesthesia; Warmed solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warmed Saline (Experimental): Patients allocated to this arm will receive a warmed (39ºC) solution of up to 500mL of isotonic saline. This solution will be administered directly to the cerebral vasculature as part of the angiography.
  Interventions: Other: Warmed Isotonic Saline
- Room-Temperature Saline (Active Comparator): Patients allocated to this arm will receive isotonic saline at room temperature. This solution will be administered directly to the cerebral vasculature as part of the angiography.
  Interventions: Other: Room-Temperature Isotonic Saline

INTERVENTIONS:
Other: Warmed Isotonic Saline — Isotonic saline warmed to 39ºC.
  Arms: Warmed Saline
Other: Room-Temperature Isotonic Saline — Isotonic saline at room temperature
  Arms: Room-Temperature Saline

SUMMARY:
This study evaluates whether the use of warmed solutions during cerebral angiography reduces the incidence of post-anaesthetic shivering. Half of participants will receive pre-warmed (39ºC) isotonic saline, while the other half receives the same solution at room temperature.

DETAILED DESCRIPTION:
Shivering is a physiologic reaction aimed at raising body temperature that is very common amongst patients undergoing cerebral angiographies. The use of pre-warmed solutions during the procedure may reduce the incidence of shivering amongst these patients. In this triple-blind randomised trial, a consecutive sample of participants receiving total intravenous anaesthesia (TIVA) and undergoing cerebral angiography will be allocated to receive a warmed (39ºC) solution of up to 500cc of isotonic saline or the same solution, but at room temperature. Patients requiring sedation, those expected to require mechanical ventilation after the procedure, those with diminished consciousness (Glasgow Coma Scale <15 pts) and patients not wishing to participate will be excluded from the study. The primary endpoint for this study is the incidence of shivering up to 60 minutes after the procedure is completed. Shivering will be assessed using a validated scale by operators unaware of treament allocation. All analyses will be undertaken by a statistician that will not participate of the clinical assessment of included patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving TIVA
* Patients undergoing cerebral angiography

Exclusion Criteria:

* Glasgow Coma Scale <15 points prior to procedure
* Expected need of mechanical ventilation after procedure completion
* Use of sedatives
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Postprocedural Shivering | up to 60 minutes
  Once the procedure is completed, the patient will be extubated and the presence or absence of shivering will be recorded up to 60 minutes after the extubation with the Badjatia 2008 scale consisting of a gradual evaluation of 0 to 3 points. With scores greater or equal to 1, shivering is considered established.

SECONDARY OUTCOMES:
Shivering severity | 60 minutes
  The post operative shivering scale of Badjatia 2008 will be used. It consist of a gradual evaluation of 0 to 3 points, with 0 being the absence of shivering, 1 slight shivering, 2 moderate and 3 severe. The highest score obtained will be recorded within the measurements made every 5 minutes in the first 60 minutes after extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Lopez, MD, Study Director — Hospital Carlos Van Buren; Alvaro Silva, MD, Principal Investigator — Universidad de Valparaiso; Felipe Martinez, M.D; M.Sc., Principal Investigator — Universidad Andrés Bello
Locations (1):
- Hospital Carlos Van Buren, Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No